CLINICAL TRIAL: NCT06316245
Title: Evaluation of Days Alive and Out of Hospital at 30 Days in Patients With Poor or Good Functional Capacity Undergoing Gastrointestinal Surgery
Brief Title: Functional Capacity and Days Alive Out of Hospital at 30 Days
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Muserref Beril Dincer, Medical Doctor, Istanbul University
Other Study IDs: 2024/178
Record Dates: First submitted 2024-02-29; First posted 2024-03-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group DASI ≤ 34: Patients with Duke Activity Status Index (DASI) scores are ≤ 34 before the surgery.
  Interventions: Other: DASI questionnaire
- Group DASI > 34: Patients with Duke Activity Status Index (DASI) scores are > 34 before the surgery.
  Interventions: Other: DASI questionnaire

INTERVENTIONS:
Other: DASI questionnaire — All patients will answer the DASI questionnaire before surgery. According to their scores, they will be divided into two groups. A score of 34 and below will be considered poor, and above 34 will be considered to have good functional capacity.

SUMMARY:
This prospective observational study aims to compare days alive and out of hospital at 30 days (DAOH-30) in patients with poor or good functional capacity undergoing gastrointestinal surgeries. The investigators are testing the hypothesis that patients with good functional capacity will have longer days alive and out of hospital than those with poor.

DETAILED DESCRIPTION:
Days Alive and Out of Hospital (DAOH) is a composite patient-centered outcome that integrates three critical clinical outcomes: death, hospital length of stay, and hospital readmission. It is associated with patient comorbidities, surgical complexity, and postoperative complications.

Evaluation of functional capacity before noncardiac surgery is recommended to identify the perioperative risks. Duke Activity Status Index (DASI) is one of the tools for determining functional capacity; the scores are between 0 and 58,2, and high scores are related to improved capacity. A DASI score of 34 and below was found to be a risk for moderate to severe complications and new disability.

The primary aim is to compare days alive and out of the hospital at 30 days in patients ≤ 34 and above 34 DASI scores. The secondary aims are to evaluate intensive care unit (ICU) need and duration, length of hospital stay, rehospitalization, postoperative complications, morbidity, and mortality in patients with DASI scores ≤ 34 and above 34. Days alive and out of hospital at 90 days will be compared in both groups as a secondary outcome. The investigators will also analyze the possible perioperative factors affecting the days alive and out of the hospital outcome.

Before the operation, the patients will answer the DASI questionnaire in the waiting area of the operating theatres. The patients will be divided into two groups according to the DASI score (Poor functional capacity: ≤ 34 points, good functional capacity: above 34 points).

Patient and surgical characteristics (comorbidities, American Society of Anesthesiologists physical status classification, laboratory values before the operation, frailty index value, American College of Surgeons Risk Calculator outcomes, surgery type, length of operation, intraoperative complications), ICU need and duration will be recorded. Postoperative complications ( cardiovascular, pulmonary, renal, neurologic, surgical, infectious, and wound ), the Postoperative Morbidity Survey (POMS) related morbidity and mortality on the 30th day will be investigated. Length of hospital stay starting with index surgery, rehospitalization and duration of further stays will be recorded. Days Alive and Out of Hospital at 30 days (DAOH-30) will be calculated using mortality, hospital length of stay, and readmissions between the date of the index surgery and the 30th postoperative day. 90th-day mortality and Days Alive and Out of Hospital at 90 days (DAOH-90) will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing intermediate and major upper or lower gastrointestinal surgeries (small intestine, colon, rectal, gastric, esophagus) with a predicted hospital stay of more than 24 hours
* Patients aged 18 and above
* Signed written informed consent
* Reaching all perioperative data

Exclusion Criteria:

* Day case/ambulatory or one overnight hospital stay for minor gastrointestinal and perianal surgeries (hernia repair, hemorrhoidectomy, perianal abscess and fistula, appendectomy)
* Hepatobiliary surgeries (hepatectomy, pancreas and gallbladder surgeries)
* Patients aged below 18
* Not signed written informed consent
* Missing perioperative data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing gastrointestinal surgeries at Istanbul Medical Faculty in Istanbul-Turkey will be selected for the study population. Istanbul Medical Faculty is a tertiary center university hospital with approximately 25.000 surgeries annually.
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-08-19 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital at 30 days (DAOH-30) | 30 days
  It is calculated using mortality, hospital length of stay, and readmissions between the date of the index surgery and the 30th postoperative day.

SECONDARY OUTCOMES:
Days alive and out of hospital at 90 days (DAOH-90) | 90 days
  It is calculated using mortality, hospital length of stay, and readmissions between the date of the index surgery and the 90th postoperative day.
Postoperative complications | 30 days
  Cardiovascular, pulmonary, renal, neurologic, surgical, infectious and wound complications
The Postoperative Morbidity Survey (POMS) defined morbidity | 30 days
  Pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, hematological, wound complications and pain will be examined according to POMS
Mortality | 30 days and 90 days
  In and out of hospital mortality
Intensive care unit (ICU) stay | 30 days
  Duration of ICU stay (days)
Length of hospital stay after index surgery | 30 days
  Length of first hospital stay starting with index surgery (days)
Rehospitalization | 30 days and 90 days
  Readmission and hospitalization after first discharge

CONTACTS AND LOCATIONS:
Overall Officials: Muserref B Dincer, Principal Investigator — Istanbul University, Istanbul Medical Faculty, Department Anesthesiology and Reanimation
Locations (1):
- Istanbul University Istanbul Medical Faculty, Department of Anesthesiology and Reanimation, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No